CLINICAL TRIAL: NCT02326324
Title: The University Hospital of South Manchester Cardiovascular Magnetic Resonance Study
Brief Title: The UHSM Cardiovascular Magnetic Resonance Study
Acronym: UHSM CMR
Status: Active, not recruiting | Type: Observational
Sponsor: Manchester University NHS Foundation Trust (Other Government)
Collaborators: University of Pittsburgh Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 14/NW/1165; 2014CD013 (Other: Manchester University NHS Foundation Trust)
Record Dates: First submitted 2014-12-22; First posted 2014-12-29 (Estimated); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral blood sampling will be performed on the same day as CMR scanning
Oversight: Data Monitoring Committee: No

SUMMARY:
This study aims to investigate the diagnostic and prognostic utility of cardiovascular magnetic resonance (CMR) imaging in a large cohort of unselected patients who are undergoing CMR scanning for clinical indications (i.e. suspected/confirmed cardiovascular disease). CMR indices will be related to the presence and severity of cardiovascular disease and other markers of cardiovascular and health status.

DETAILED DESCRIPTION:
Patients will undergo CMR scanning in the usual clinical manner. As part of the study, patients will undergo approximately 5 minutes of extra CMR scanning. Cardiovascular anatomical, structural and functional data will be recorded, including data pertaining to myocardial characteristics (e.g. extracellular volume, oedema, fibrosis, infarction, function, perfusion), pericardial disease; valvular disease; vascular structure and function.

Blood sampling will be performed on the same day as CMR scanning for assessment of serum/plasma markers of cardiovascular disease and health status, and DNA analysis. Health questionnaires will be completed on the day of CMR scanning.

Follow-up information regarding health status, demographics and concurrent medical conditions and treatments will be obtained over a 10 year period following CMR scanning.

ELIGIBILITY:
Inclusion Criteria:

Any adult patient undergoing clinically indicated CMR scanning at the UHSM CMR Unit.

Exclusion Criteria:

Age < 18 years, imprisonment, inability to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients undergoing clinically indicated CMR scanning (i.e. patients with suspected or confirmed cardiovascular disease)
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2015-01-05 (Actual); Primary Completion 2029-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
All cause mortality | 10 years with planned interim analyses

SECONDARY OUTCOMES:
Cardiovascular death | 10 years with planned interim analyses
Hospitalisation for heart failure | 10 years with planned interim analyses
Development of cardiovascular disease | 10 years with planned interim analyses
Development of complications of cardiovascular disease | 10 years with planned interim analyses

CONTACTS AND LOCATIONS:
Overall Officials: Christopher A Miller, MBChB, PhD, Principal Investigator — University Hospital of South Manchester; Matthias Schmitt, MD, PhD, Principal Investigator — University Hospital of South Manchester
Locations (1):
- University Hospital of South Manchester, Manchester, Greater Manchester, United Kingdom

REFERENCES:
- [Derived] Bradley J, Schelbert EB, Bonnett LJ, Lewis GA, Lagan J, Orsborne C, Brown PF, Black N, Naish JH, Williams SG, McDonagh T, Schmitt M, Miller CA. Growth differentiation factor-15 in patients with or at risk of heart failure but before first hospitalisation. Heart. 2024 Jan 10;110(3):195-201. doi: 10.1136/heartjnl-2023-322857. PMID 37567614
- [Derived] Di Marco A, Brown PF, Bradley J, Nucifora G, Anguera I, Miller CA, Schmitt M. Extracellular volume fraction improves risk-stratification for ventricular arrhythmias and sudden death in non-ischaemic cardiomyopathy. Eur Heart J Cardiovasc Imaging. 2023 Mar 21;24(4):512-521. doi: 10.1093/ehjci/jeac142. PMID 35877070